CLINICAL TRIAL: NCT04602273
Title: Treatment of High Risk Myelodysplastic Syndromes (MDS) Not Candidates for Allogeneic Transplantation of Hematopoietic Progenitors (ALO-HSCT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Collaborators: Hospital Son Llatzer (Other); Germans Trias i Pujol Hospital (Other); Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CET-AZA-2016-01
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 ml Bone Marrow Aspirate samples will be processed and stored at: Laboratorio de Hematología Primera Planta Edificio General ICO - Hospital Germans Trias i Pujol Ctra. Canyet s/n 08916 Badalona
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High Risk MDS: New diagnosed patients treated with Azacitidine 75 mg/sqm SC QD on a 28 days based cycles (both 7-0-0 and 5-0-2 regimens are allowed) until disease progression, unacceptable toxicity, death or investigator decision
  Interventions: Drug: Azacitidine Injection [Vidaza]

INTERVENTIONS:
Drug: Azacitidine Injection [Vidaza]

SUMMARY:
An observational, non-interventional, prospective and multicenter study of Azacitidine in newly diagnosed High Risk Myelodysplastic Syndromes.

Primary objectives are to asses mutational status of target genes by Next Generation Sequencing, to evaluate prognostic value of geriatric assessment scales and to evaluate overall survival.

The main hypothesis is that mutation status of target genes and geriatric scales have statistical significant impact on overall survival.

Study time points will be at diagnosis, 6, 12, 18 and 24 months, always taking into account the routine clinical practice, when sample to assess mutational status will be collected. Geriatric assessment will only be performed at diagnosis.

Upon the signature of informed consent and the checking of inclusion criteria, patients will receive treatment with Azacitidine 75 mg/sqm on a 28 days based cycles (both 7-0-0 and 5-0-2 regimens are allowed) until disease progression, unacceptable toxicity or investigator decision.

150 patients are expected to be recruited at study sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with myelodysplastic syndrome (MDS) according to WHO criteria, including non-proliferative chronic myelomonocytic leukemia (CMML) that is considered high risk, and not candidates for transplantation.
* High-risk MDS: (following the Grupo Español Síndrome Mielodisplásico, GESDM MDS guides) and the recommendations of Valcárcel, D. et al).

Median expected OS less than 30 months. Intermediate-2 or high risk IPSS and / or high or very high risk WPSS and / or high or very high risk IPSSS-R.

IPSS of intermediate risk and / or WPSS of intermediate risk and / or IPSS-R of intermediate risk that present at least one of the following characteristics:

Cytogenetic abnormality of the IPSS-R high or very high cytogenetic risk group Platelet count <30 x10E9/l Neutrophil count <0.5 x 10E9 / l Presence of dense and diffuse myelofibrosis, with or without collagen formation (grades 2-3 of the European consensus) Category 3 of the LRSS score (MD Anderson low risk score system)

* Patient diagnosed with LAM de novo according to WHO criteria, with 20-30% blasts count in bone marrow, trilineal dysplasia and more than 70 years and not candidate for intensive chemotherapy.
* Willing to provide voluntary written informed consent

Exclusion Criteria:

* Serious active medical condition, not related to MDS, that could limit patient compliance and follow-up or that, in the Investigator's opinion,could compromise the patient's safety.
* Presence of other active malignant disease
* Organic function parameters: (except when the alteration is due to MDS) Hepatic: Bilirubin> 2 x upper limit of normal (ULN) Renal: Creatinine> 2 x upper limit of normal (ULN)
* Ejection fraction (<40%) and / or symptomatic heart failure.
* Leukaemia secondary to Myeloproliferative Syndrome.
* Serious psychiatric or neurological disease.
* Positive Serology for HIV.
* Proliferative CMML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed High-Risk Myelodysplastic Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5- year overall survival
Progression Free Survival (PFS) | 5-year progression free survival
Overall Response Rate (OOR) | 12 months OOR
Treatment-Emergent Adverse Events Rate (TEAE) | 12 Months TEAE rate

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bargay, MD PhD, Principal Investigator — Hospital Son Llatzer; Lurdes Zamora, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Son Llàtzer, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided
There is not a confirmed IPD sharing plan. It will be confirmed by Principal Investigators

REFERENCES:
- [Background] Tefferi A, Vardiman JW. Myelodysplastic syndromes. N Engl J Med. 2009 Nov 5;361(19):1872-85. doi: 10.1056/NEJMra0902908. No abstract available. PMID 19890130
- [Background] Germing U, Strupp C, Kundgen A, Bowen D, Aul C, Haas R, Gattermann N. No increase in age-specific incidence of myelodysplastic syndromes. Haematologica. 2004 Aug;89(8):905-10. PMID 15339672
- [Background] Cazzola M, Malcovati L. Myelodysplastic syndromes--coping with ineffective hematopoiesis. N Engl J Med. 2005 Feb 10;352(6):536-8. doi: 10.1056/NEJMp048266. No abstract available. PMID 15703418
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Fega KR, Abel GA, Motyckova G, Sherman AE, DeAngelo DJ, Steensma DP, Galinsky I, Wadleigh M, Stone RM, Driver JA. Non-hematologic predictors of mortality improve the prognostic value of the international prognostic scoring system for MDS in older adults. J Geriatr Oncol. 2015 Jul;6(4):288-98. doi: 10.1016/j.jgo.2015.05.003. Epub 2015 Jun 11. PMID 26073533
- [Background] Hamaker ME, Mitrovic M, Stauder R. The G8 screening tool detects relevant geriatric impairments and predicts survival in elderly patients with a haematological malignancy. Ann Hematol. 2014 Jun;93(6):1031-40. doi: 10.1007/s00277-013-2001-0. Epub 2014 Feb 2. PMID 24488257
- [Background] Bonanad S, De la Rubia J, Gironella M, Perez Persona E, Gonzalez B, Fernandez Lago C, Arnan M, Zudaire M, Hernandez Rivas JA, Soler A, Marrero C, Olivier C, Altes A, Valcarcel D, Hernandez MT, Oiartzabal I, Fernandez Ordono R, Arnao M, Esquerra A, Sarra J, Gonzalez-Barca E, Gonzalez J, Calvo X, Nomdedeu M, Garcia Guinon A, Ramirez Payer A, Casado A, Lopez S, Duran M, Marcos M, Cruz-Jentoft AJ; GAH Group. Development and psychometric validation of a brief comprehensive health status assessment scale in older patients with hematological malignancies: The GAH Scale. J Geriatr Oncol. 2015 Sep;6(5):353-61. doi: 10.1016/j.jgo.2015.03.003. Epub 2015 Jun 29. PMID 26139300
- [Background] Rollison DE, Howlader N, Smith MT, Strom SS, Merritt WD, Ries LA, Edwards BK, List AF. Epidemiology of myelodysplastic syndromes and chronic myeloproliferative disorders in the United States, 2001-2004, using data from the NAACCR and SEER programs. Blood. 2008 Jul 1;112(1):45-52. doi: 10.1182/blood-2008-01-134858. Epub 2008 Apr 28. PMID 18443215
- [Background] Klepin HD. Myelodysplastic Syndromes and Acute Myeloid Leukemia in the Elderly. Clin Geriatr Med. 2016 Feb;32(1):155-73. doi: 10.1016/j.cger.2015.08.010. PMID 26614866
- [Background] Xicoy B, Jimenez MJ, Garcia O, Bargay J, Martinez-Robles V, Brunet S, Arilla MJ, Perez de Oteyza J, Andreu R, Casano FJ, Cervero CJ, Bailen A, Diez M, Gonzalez B, Vicente AI, Pedro C, Bernal T, Luno E, Cedena MT, Palomera L, Simiele A, Calvo JM, Marco V, Gomez E, Gomez M, Gallardo D, Munoz J, de Paz R, Grau J, Ribera JM, Benlloch LE, Sanz G. Results of treatment with azacitidine in patients aged >/= 75 years included in the Spanish Registry of Myelodysplastic Syndromes. Leuk Lymphoma. 2014 Jun;55(6):1300-3. doi: 10.3109/10428194.2013.834532. Epub 2013 Sep 16. PMID 23952246
- [Background] Gangat N, Patnaik MM, Tefferi A. Myelodysplastic syndromes: Contemporary review and how we treat. Am J Hematol. 2016 Jan;91(1):76-89. doi: 10.1002/ajh.24253. PMID 26769228
- [Background] Bejar R, Lord A, Stevenson K, Bar-Natan M, Perez-Ladaga A, Zaneveld J, Wang H, Caughey B, Stojanov P, Getz G, Garcia-Manero G, Kantarjian H, Chen R, Stone RM, Neuberg D, Steensma DP, Ebert BL. TET2 mutations predict response to hypomethylating agents in myelodysplastic syndrome patients. Blood. 2014 Oct 23;124(17):2705-12. doi: 10.1182/blood-2014-06-582809. Epub 2014 Sep 15. PMID 25224413
- [Background] Itzykson R, Kosmider O, Cluzeau T, Mansat-De Mas V, Dreyfus F, Beyne-Rauzy O, Quesnel B, Vey N, Gelsi-Boyer V, Raynaud S, Preudhomme C, Ades L, Fenaux P, Fontenay M; Groupe Francophone des Myelodysplasies (GFM). Impact of TET2 mutations on response rate to azacitidine in myelodysplastic syndromes and low blast count acute myeloid leukemias. Leukemia. 2011 Jul;25(7):1147-52. doi: 10.1038/leu.2011.71. Epub 2011 Apr 15. PMID 21494260
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Deschler B, Ihorst G, Platzbecker U, Germing U, Marz E, de Figuerido M, Fritzsche K, Haas P, Salih HR, Giagounidis A, Selleslag D, Labar B, de Witte T, Wijermans P, Lubbert M. Parameters detected by geriatric and quality of life assessment in 195 older patients with myelodysplastic syndromes and acute myeloid leukemia are highly predictive for outcome. Haematologica. 2013 Feb;98(2):208-16. doi: 10.3324/haematol.2012.067892. Epub 2012 Aug 8. PMID 22875615
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- See also: Grupo Español de Sindrome Mielodiplásico (GESMD) MDS treatment guides — https://gesmd.es/pdfs/guias_smd/Haematologia_Guias_SMD.pdf